CLINICAL TRIAL: NCT03437044
Title: A Randomized Comparison of Platelet Inhibition Using a Low Maintenance Dose Ticagrelor Regimen Versus Standard Dose Clopidogrel in Diabetes Mellitus Patients Without Prior Major Cardiovascular Events Undergoing Elective Percutaneous Coronary Intervention: The OPTIMUS (Optimizing Antiplatelet Therapy in Diabetes Mellitus)-6 Study
Brief Title: Low Maintenance Dose Ticagrelor Versus Clopidogrel in Diabetes Patients Undergoing PCI
Acronym: OPTIMUS-6
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR 13396
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Artery Disease
Keywords: diabetes mellitus; percutaneous coronary intervention; ticagrelor; clopidogrel; coronary artery disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Diabetes Mellitus | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Intervention Model Description: Prospective randomized
Masking Description: Staff performing PK/PD assessments will remain blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ticagrelor (Experimental): 180 mg loading dose (LD) followed by a 60 mg bid maintenance (MD) starting 12 h (± 1 h) after the LD
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): 600 mg LD followed by a 75 mg od MD starting 24 hours (± 1 h) after the LD
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — After providing written informed consent and following diagnostic angiography, patients meeting study entry criteria undergoing PCI will be randomly assigned in a 1:1 ratio to treatment with either ticagrelor or clopidogrel. Randomized treatment will be maintained for 30±3 days.
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Clopidogrel — After providing written informed consent and following diagnostic angiography, patients meeting study entry criteria undergoing PCI will be randomly assigned in a 1:1 ratio to treatment with either ticagrelor or clopidogrel. Randomized treatment will be maintained for 30±3 days.
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
To date there is very little PD and pharmacokinetic (PK) data on the ticagrelor 60 mg bid dosing regimen. In particular, there is no prospective PK/PD study on this dosing regimen in patients with DM who are known to have impaired response to clopidogrel therapy. Since DM patients frequently require elective PCI due to chronic progression of CAD (and not solely because of an acute thrombotic complication), and clopidogrel remains the guideline recommended P2Y12 inhibiting therapy for these patients, understanding the PD effects of the ticagrelor 60 mg bid regimen in this setting is an unmet clinical need. This is also in light of the ongoing THEMIS trial which is specifically evaluating the impact of the ticagrelor 60 mg bid dosing regimen in type 2 DM patients without a prior major CV event.

DETAILED DESCRIPTION:
Patients with diabetes mellitus (DM) are characterized by platelet hyperreactivity and reduced pharmacodynamic (PD) effects to several oral antiplatelet agents, including clopidogrel. In addition to the hyperreactive platelet phenotype, impaired drug metabolism as well as increased platelet turnover rates may contributed to impaired clopidogrel-induced antiplatelet effects in DM patients. These observations may contribute to the higher ischemic event rates, including stent thrombosis, observed in DM patients compared with non-DM patients treated with clopidogrel.

Ticagrelor is characterized by more prompt, potent and predictable antiplatelet effects compared with clopidogrel and lower ischemic events in patients with an acute coronary syndrome (ACS) on a background of aspirin therapy. In patients who experienced a prior (1-3 years) myocardial infarction (MI), compared with placebo, ticagrelor 60 mg bid on a background of aspirin therapy also reduced long-term ischemic events, with a mortality benefit observed in DM patients.

To date the PD effects of ticagrelor versus clopidogrel in DM largely derive from post-hoc assessments or in stabilized patients (e.g. >30 days after PCI), and have not been prospectively evaluated in the context of elective PCI procedures. Moreover, PD studies with the ticagrelor 60 mg bid regimen are limited. Therefore, the aim of this investigation will be to compare the PD effects of a ticagrelor 60 mg bid versus clopidogrel 75 mg od MD regimen in DM patients without a prior major CV event undergoing elective PCI.

ELIGIBILITY:
Inclusion criteria:

1. Provision of informed consent prior to any study specific procedures
2. Men or women ≥18 years of age
3. Diagnosed with type 2 DM defined by ongoing glucose lowering drug (oral medications and / or insulin) treatment for at least 1 month
4. Presence of CAD undergoing elective PCI* * Patients will need to be cardiac enzyme-negative prior to undergoing coronary angiography. Patient will need to be on a background of aspirin therapy (treated with a 325 mg LD prior to coronary angiography unless already on chronic low-dose aspirin therapy). Patients on maintenance clopidogrel 75 mg therapy for at least 1 week due to a prior vascular intervention will also be eligible. However, patients on clopidogrel, ticagrelor or prasugrel due to a prior acute major cardiovascular event (MI or stroke) will not be eligible.

Exclusion criteria:

1. Previous MI (with the exception of definite non-type 1 MI [eg, due to coronary revascularization procedure, profound hypotension, hypertensive emergency, tachycardia, or profound anemia])
2. Previous stroke (transient ischemic attack [TIA] is not included in the stroke definition)
3. Use of an intravenous antiplatelet therapy (i.e., cangrelor or GPI) during PCI
4. On treatment with clopidogrel, prasugrel, or ticagrelor due to a prior acute major CV event (MI or stroke) (on treatment with clopidogrel due to prior vascular intervention not secondary to a major CV event is allowed)
5. Planned use of aspirin treatment at doses >100 mg od
6. Anticipated concomitant oral or intravenous therapy with strong cytochrome P450 3A4 (CYP3A4) inhibitors or CYP3A4 substrates with narrow therapeutic indices that cannot be stopped for the course of the study:

   * Strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin (but not erythromycin or azithromycin), nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atanazavir
   * CYP3A4 substrates with narrow therapeutic index: quinidine, simvastatin at doses >40 mg daily or lovastatin at doses >40 mg daily
7. Need for chronic oral anticoagulant therapy or chronic low-molecular-weight heparin (at venous thrombosis treatment not prophylaxis doses)
8. Patients with known bleeding diathesis or coagulation disorder
9. History of previous intracerebral bleed at any time, gastrointestinal (GI) bleed within the past 6 months prior to randomization, or major surgery within 30 days prior to randomization
10. Active pathological bleeding
11. Hypersensitivity to ticagrelor and clopidogrel or any of the excipients
12. Increased risk of bradycardic events (eg, known sick sinus syndrome, second or third degree AV block or previous documented syncope suspected to be due to bradycardia) unless treated with a pacemaker
13. Known severe liver disease (eg, ascites and/or clinical signs of coagulopathy)
14. Renal failure requiring dialysis
15. Known platelet count <80x106/mL
16. Known hemoglobin <9 g/dL
17. Women of child-bearing potential (ie, those who are not chemically or surgically sterilized or who are not post-menopause) who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator OR who have a positive pregnancy test at enrolment or randomization OR women who are breast-feeding. If a subject becomes pregnant during the course of the study the investigational product should be discontinued immediately [the outcome of all pregnancies (spontaneous miscarriage, elective termination, ectopic pregnancy, normal birth or congenital abnormality) will be followed up and documented even if the subject was discontinued from the study].
18. Inability of the patient to understand and/or comply with study procedures and/or follow up, in the opinion of the investigator, OR any conditions that, in the opinion of the investigator, may render the patient unable to complete the study
19. Life expectancy of less than 1 month based on investigator's judgement
20. Participation in another clinical study with an investigational (defined as non-FDA approved) product within 28 days prior to enrolment
21. Previous randomization in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2020-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD,PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ticagrelor | Clopidogrel
Started | 20 | 20
Completed | 17 | 18
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Clopidogrel | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7) | 66 (9) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 12 | 17 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: P2Y12 Reaction Units (PRU)
Description: The primary endpoint of our study will be platelet reactivity, measured as PRU level using VerifyNow PRU, of ticagrelor versus clopidogrel MD at 30 days after PCI, immediately pre-dosing dosing (trough levels). PRU is a marker of platelet reactivity. Higher PRU values correspond to higher aggregation and lower response to antiplatelet therapy.
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: PRU
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 17 | 18
PRU | 60 [32 to 89] | 146 [106 to 185]
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Test type: Superiority; p = 0.001, ANCOVA; the corresponding baseline value of platelet reactivity was used as covariate

2. Secondary Outcome: Platelet Reactivity Index (PRI)
Description: Platelet reactivity measured as PRI% using whole blood vasodilator-stimulated phosphoprotein (VASP), of ticagrelor versus clopidogrel MD at 30 days after PCI, immediately pre-dosing dosing (trough levels). PRI% is a marker of platelet reactivity. Higher PRI values correspond to higher aggregation and lower response to antiplatelet therapy.
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: PRI %
Arm/Group | Ticagrelor | Clopidogrel
Number analyzed (Participants) | 17 | 18
PRI % | 25 [14 to 35] | 65 [55 to 76]
Statistical Analysis 1: Comparison: Ticagrelor vs Clopidogrel; Test type: Superiority; p < 0.001, ANCOVA; the corresponding baseline value of platelet reactivity was used as covariate

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Ticagrelor | Clopidogrel
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=20) | Clopidogrel (N=20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT03437044/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT03437044/ICF_001.pdf